CLINICAL TRIAL: NCT00132574
Title: Milk Minimization and Acne Recurrence Trial (MMART)
Brief Title: Pilot Study of a Dietary Intervention to Prevent Acne Recurrence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Department of Dermatology, Leeds General Infirmary (Unknown); Breast Cancer Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BCRF-P11733; SRC200402
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2006-09-21 (Estimated); Status verified 2006-09

CONDITIONS: Acne
Keywords: acne, dairy
MeSH Terms: conditions — Acne Vulgaris | interventions — Dairy Products

INTERVENTIONS:
Behavioral: Minimization of milk and dairy products in the diet

SUMMARY:
The purpose of this study is to determine whether minimizing the intake of milk and dairy products will reduce the recurrence of acne among people who have been successfully treated for acne with isotretinoin.

DETAILED DESCRIPTION:
Acne is one of the most common dermatologic diseases affecting 40 to 50 million people in the United States, most of who are adolescents and young adults. In addition to the well-recognized physical sequelae of this condition, several studies have linked severe acne to considerable social impairments and serious psychological conditions including suicidal ideation and major depression. Furthermore, severe acne has been recognized in some studies as a risk factor for breast cancer, suggesting that these conditions may have common causes. Little is known about the role of diet in the pathogenesis of acne. Recent analyses of the Nurses' Health Study II and the Growing-Up Today Study suggest that high intake of milk increases the risk of developing acne during adolescence. Despite the consistency of findings between these two studies, they cannot be regarded as conclusive and further research is needed in this area. Establishing the nature of the association between milk intake and acne can have broad clinical and public health implications. It could enhance the currently existing therapeutic options for the treatment of acne. More importantly, public health recommendations regarding milk and dairy intake could be designed in order to prevent its effects on the sebaceous glands and probably other hormone sensitive glands like the breast.

To test the hypothesis that milk intake increases the risk of developing acne, we will compare the effect of minimizing milk and dairy intake against not making changes in the diet of subjects who usually consume at least 2 servings/day of milk and dairy products on the recurrence of acne lesions among patients previously treated with isotretinoin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 16 and 25 years of age who have successfully completed treatment for acne with oral isotretinoin.
* Patients who regularly consume at least 2 servings (480ml) of milk per day.
* Patients who can attend scheduled study follow-up visits at the Leeds General Infirmary.
* Patients who grant informed consent for participation in the study.
* Patients who agree to comply with the intervention and follow-up procedures in the study.

Exclusion Criteria:

* Patients who received isotretinoin for a condition other than acne (e.g Malassezia folliculitis).
* Patients who have been off isotretinoin for more than 60 days at the moment of enrolment into the study.
* Patients who used any topical or oral acne medications between the end of therapy with isotretinoin and enrolment in the study.
* Patients who have been previously diagnosed with an endocrinologic disorder likely to cause acne such as polycystic ovary syndrome, congenital adrenal hyperplasia, adrenal or ovarian tumors or any other hyperandrogenemic states.
* Patients who are using any of the following medications which are likely to cause or abate acne:

  * Corticosteroids;
  * Contraceptives containing medroxyprogesterone acetate, norgestrel or levonorgestrel;
  * Dilantin or other antiepileptic;
  * Finasteride, spironolactone or flutamide;
  * Testosterone or dietary body-building protein powders.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2005-08; Study Completion 2006-09

PRIMARY OUTCOMES:
Number of recurrent acne lesions

SECONDARY OUTCOMES:
Time to re-initiation of treatment for acne

CONTACTS AND LOCATIONS:
Overall Officials: Walter C Willett, MD, DrPH, Principal Investigator — Harvard School of Public Health (HSPH); Jorge E Chavarro, MD, SM, Study Director — Harvard School of Public Health (HSPH); F. William Danby, MD, FRCPC, Study Director
Locations (1):
- Department of Dermatology, Leeds General Infirmary, Leeds, United Kingdom